CLINICAL TRIAL: NCT03562026
Title: Specific Clinical Experience Investigation of Nexium in Paediatric Patients
Brief Title: S-CEI of Nexium in Paediatric Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961WC00002
Record Dates: First submitted 2018-04-29; First posted 2018-06-19 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Peptic Ulcer, Gastroesophageal Reflux
MeSH Terms: conditions — Peptic Ulcer; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To capture safety and efficacy when Nexium are administered to pediatric patients in clinical practice after launch

DETAILED DESCRIPTION:
The objective of this investigation is to capture the followings when Nexium capsules or Nexium granules for suspension (single-dose package) are administered to pediatric patients in clinical practice after launch.

1. Development of adverse reactions which are unexpected from Precaution for Use
2. Development of adverse reactions
3. Efficacy

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1(inclusive) to 15 (exclusive) years
* Patients who have been prescribed Nexium for the first time for "gastric ulcer", "duodenal ulcer", "anastomotic ulcer", "reflux oesophagitis", "non-erosive reflux disease", or "Zollinger-Ellison syndrome", .

Exclusion Criteria:

* Patients with a history of hypersensitivity to components contained in this product.
* Patients during treatment with Atazanavir Sulfate and Rilpivirine hydrochloride.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 1(inclusive) to 15 (exclusive) years and who have been prescribed Nexium for the first time for "gastric ulcer", "duodenal ulcer", "anastomotic ulcer", "reflux oesophagitis", "non-erosive reflux disease", or "Zollinger-Ellison syndrome", which are the indications of Nexium.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
frequency of adverse drug reactions (ADRs) | up to 8 weeks
  Development of ADRs by unexpected from "Precautions for Use" of Nexium JPI, by SOC, by patient demography and by treatment
rate of improvement/worsening of symptoms | up to 8 weeks
  Rage of improvement/worsening of symptoms and cure rate on endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Toshihito Nakano, Study Director — AZKK
Locations (31):
- Japan (31):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Numakunai
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Toyama
  - Research Site, Yamagata

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D961WC00002&attachmentIdentifier=361f2d48-69fa-4d2c-a1ae-ae84372cb1db&fileName=CSR_cynopsis_D961WC00002.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D961WC00002&attachmentIdentifier=c793c729-36ad-4130-bd26-823ddb0cabac&fileName=JP_PMS_Protocol_NEX_D961WC00002_E_redacted.pdf&versionIdentifier=